CLINICAL TRIAL: NCT04905563
Title: Post-operative Pain Management in Supracondylar Humerus Fractures: A Randomized, Double-blinded, Prospective Study
Brief Title: NSAIDs vs Opioids for Post-op Pain in Supracondylar Humerus Fractures
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Clinical evidence supporting the hypothesis of this study has been published
Sponsor: Le Bonheur Children's Hospital (Other)
Collaborators: The Campbell Foundation (Other)
Responsible Party: Principal Investigator, Lindsey Locke, Pediatric Nurse Practitioner, Le Bonheur Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Post-op SCHF Pain
Record Dates: First submitted 2021-05-21; First posted 2021-05-27 (Actual); Results first posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Supracondylar Humerus Fracture
Keywords: Elbow surgery; Pain
MeSH Terms: conditions — Pain | interventions — oxycodone-acetaminophen; Acetaminophen; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (Other): Standard of care- weight based dose of liquid acetaminophen-hydrocodone- 0.15 mg/kg/dose every six hours with a max dose of 10 mg/dose
  Interventions: Drug: Acetaminophen-Hydrocodone
- Treatment (Experimental): Weight based dose of liquid acetaminophen and ibuprofen- acetaminophen 15 mg/kg/dose and ibuprofen 10 mg/kg/dose every six hours with a max dose of 650 mg/dose of acetaminophen and 600 mg/dose of ibuprofen.
  Interventions: Drug: Acetaminophen and Ibuprofen

INTERVENTIONS:
Drug: Acetaminophen-Hydrocodone — Narcotic
  Other Names: Lortab
  Arms: Control
Drug: Acetaminophen and Ibuprofen — Non-narcotic
  Other Names: Tylenol and Advil
  Arms: Treatment

SUMMARY:
The purpose of this study is to determine if using the combination of acetaminophen (also known as Tylenol) and ibuprofen (also known as Motrin or Advil) will provide equal or better pain control as compared to acetaminophen-hydrocodone (also known as Lortab), in children with broken elbows who need surgery. This study will examine whether the combination of acetaminophen and ibuprofen can provide pain control as well as or better than acetaminophen-hydrocodone so that doctors might be able to prescribe less acetaminophen-hydrocodone (which can be addictive) to children in the future. Currently, the standard of care for pain control following this kind of elbow surgery is acetaminophen-hydrocodone.

DETAILED DESCRIPTION:
For this study, participants will be randomized (randomly assigned) to either receive scheduled acetaminophen-hydrocodone (which is the current standard of care treatment) or acetaminophen and ibuprofen (the experimental treatment) for post operative pain control following surgery for supracondylar humerus fracture. Patients in the experimental treatment group who require 2 doses of breakthrough pain medication in a row in order to control their pain will be switched to the standard of care treatment. Follow up information regarding outcomes post-discharge will be collected via secure email or text 48-72 hours post-discharge.

ELIGIBILITY:
Inclusion Criteria:

* isolated supracondylar humerus fracture
* undergoing closed reduction with percutaneous pinning (CRPP)

Exclusion Criteria:

* Allergies to acetaminophen, ibuprofen, and/or acetaminophen-HYDROcodone
* Liver or renal disease
* history of bleeding disorder
* medical diagnosis of juvenile arthritis
* on chronic NSAIDs or Opioids PRIOR to the procedure
* medical diagnosis of coagulopathies, open fractures, other injuries at time of diagnosis (multi-system trauma)
* vascular compromise and/or compartment syndrome upon admission

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Locke, MSN, Principal Investigator — Le Bonheur Children's Hospital
Locations (1):
- Le Bonheur Children's Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
No Plan has been made for such data sharing

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Treatment
Started | 15 | 15
Completed | 13 | 13
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Standard of care orders entered by resident | 1 | 0
Not completed — Patient discharged from PACU. No study meds adinistered | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Treatment | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: Years] | 6.8 (1.6) | 6.6 (0.92) | 6.7 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 8 | 7 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 3 | 2 | 5
  Hispanic | 1 | 0 | 1
  Caucasian | 9 | 11 | 20
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores
Description: Pain scores during postoperative hospital stay on a Wong-Baker Faces scale. 0 (No Pain) to 10 (Worst pain).
Time Frame: 24 hours (duration of post-operative stay)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Treatment
Number analyzed (Participants) | 13 | 13
score on a scale | 0.95 (1.35) | 0.97 (1.53)

ADVERSE EVENTS:
Time Frame: 24 hours (duration of post-operative stay)
Arm/Group | Control | Treatment
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-05): https://cdn.clinicaltrials.gov/large-docs/63/NCT04905563/Prot_SAP_002.pdf
  • Informed Consent Form (2023-08-07): https://cdn.clinicaltrials.gov/large-docs/63/NCT04905563/ICF_001.pdf